CLINICAL TRIAL: NCT04378959
Title: Randomized, Placebo-controlled Crossover Trial Evaluating Topical Lidocaine Patch(es) for Mechanical Neck Pain.
Brief Title: Lidocaine Patch for Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Pain Management Institute Bethesda-Washington-Maryland (Unknown); Walter Reed National Military Medical Center (U.S. Federal Agency); Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00233514
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Neck Pain; Neck Pain, Posterior
Keywords: Cervicalgia; Neck pain; Lidocaine; Topical
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: 4 week treatment periods, separated by a 1 to 3 week washout period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical lidocaine and placebo patches will be provided to research pharmacies at participating sites, along with site-specific randomization tables. Care providers, investigators, patients and outcome assessors will all be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine patch first (Experimental): This group will receive up to 3 lidocaine patches for 4 weeks, followed by placebo patches after a 1-3 week washout period.
  Interventions: Drug: Lidocaine patch; Drug: Placebo patch
- Placebo patch first (Placebo Comparator): This group will receive up to 3 placebo patches for 4 weeks, followed by lidocaine patches after a 1-3 week washout period.
  Interventions: Drug: Lidocaine patch; Drug: Placebo patch

INTERVENTIONS:
Drug: Lidocaine patch — Up to 3 patches will be applied for 12 hours on (e.g. from 8 AM to 8 PM for those whose pain is worse during the day, or from 8 PM to 8 AM for those whose pain is worse at night) and 12 hours off x 4 weeks.
Drug: Placebo patch — Up to 3 patches will be applied for 12 hours on (e.g. from 8 AM to 8 PM for those whose pain is worse during the day, or from 8 PM to 8 AM for those whose pain is worse at night) and 12 hours off x 4 weeks.

SUMMARY:
In this randomized, double-blind, placebo-controlled crossover study, up to 84 patients with non-radicular neck pain will be allocated in a 1:1 ratio to receive up to 3 topical lidocaine or placebo patches, to be applied 12 hours per day. At the end of 4 weeks, patients will return for patients' post-phase I treatment evaluation. Patients will crossover to receive up to 3 identical-looking topical patches of the treatment patients did not receive, to be applied in the same fashion for the same 4-week period. The primary outcome measure will be average neck pain over the past week, 4 weeks post-treatment. A positive categorical outcome (i.e. responder) will be defined as a 2-point or greater decrease in average neck pain coupled with a patient global impression of change score >/= 5/7.

DETAILED DESCRIPTION:
84 patients will be allocated to receive lidocaine patch or an identical placebo patch for phase I of this crossover study. Depending on the area of pain, up to 3 patches can be applied. Patches will be applied for 12 hours on and 12 hours off (e.g. from 8 PM to 8 AM or 8 AM to 8PM) depending on whether a person's pain is worse in the day or night.

At the end of 4 weeks of treatment, patients will return to clinic for the post-phase I treatment evaluation, at which time outcome measures will be collected. Patients will then enter a 1-week washout period, after which patients will return between 1 and 3 weeks (depending on patients' availability) to receive the treatment patch patients did not receive in phase I (i.e. lidocaine for group II patients and placebo for group I patients). The short washout period is justifiable based on the short half-life of lidocaine (90-120 minutes) and is consistent with previous topical lidocaine crossover studies. The crossover patch will be applied in the same fashion as in the 1st phase, again for a 4-week duration.

In order to reduce confounding variables, subjects in both groups must agree to not seek any additional pain management treatment as long as patients remain in the study. However, some treatments, such as physical therapy or exercise that are widely recommended can continue, so patients will be told to advise patients' pain clinic physician of any new treatments patients wish to seek during this time period. Subjects will be also be advised that patients can be prescribed rescue medications in the form of a non-steroidal anti-inflammatory drug or acetaminophen, or tramadol (up to 100 mg/d) for those who have already failed a non-steroidal anti-inflammatory drug and acetaminophen, or cannot take the drugs for medical reasons (e.g. renal disease, high cardiovascular risk).

The primary outcome measure will be average neck pain over the past week, 4 weeks post-treatment. A positive categorical outcome (i.e. responder) will be defined as a 2-point or greater decrease in average neck pain coupled with a patient global impression of change score </= 3/7.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years
* Tenderness to palpation over affected areas (using average 4 kg force for 70 kg person)
* Average pain score >/= 4 over the week prior to enrollment
* On stable doses of analgesics for 2 weeks prior to enrollment
* Chronic mechanical neck pain > 3 months in duration
* Boundaries are upper trapezius, mastoid processes, shoulders

Exclusion Criteria:

* Radicular pain as determined by clinical presentation
* Opioid dose in oral morphine equivalents/day > 30
* Moderate or severe hepatic disease (will obtain blood work and exclude individuals with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the normal range.
* Previous neck surgery
* Known structural defect presumed to be the primary pain generator (e.g. severe degenerative disc or facet joint disease)
* Serious medical (e.g. unstable angina) or psychiatric (e.g. poorly controlled depression, active substance abuse) that could interfere with treatment or pain response
* Secondary gain
* Pregnancy or breastfeeding
* painDETECT score > 18
* Known allergy to lidocaine
* Diffuse pain phenotype (e.g. fibromyalgia)
* Cervical pain greater in area than 3 patches (10 x 14 cm/patch)
* Skin defects (e.g. burns, active infection) in area(s) of application that could result in significant systemic absorption

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Mean reduction in average neck pain score on 0-10 numerical rating scale | 4 weeks
  Mean reduction in average neck pain score over the past week at week 4 compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain)

SECONDARY OUTCOMES:
Average neck pain score on 0-10 numerical rating scale | 4 weeks
  Average neck pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain)
Mean reduction in worst neck pain score on 0-10 numerical rating scale | 4 weeks
  Mean reduction in worst neck pain score over the past week at week 4 compared to baseline on 0-10 numerical rating scale (higher pain scores represent greater pain)
Worst neck pain score on 0-10 numerical rating scale | 4 weeks
  Worst neck pain score over the past week on 0-10 numerical rating scale (higher pain scores represent greater pain)
Neck disability index score | 4 weeks
  Neck disability index score on 0 to 100 percent scale (higher scores represent greater disability)
Mean reduction in neck disability index score | 4 weeks
  Mean reduction in neck disability index score over the past week at week 4 compared to baseline (higher scores represent greater disability)
Number of participants with a positive outcome | 4 weeks
  Positive outcome is defined as a greater than or equal to 2-point decrease in average neck pain on 0-10 NRS scale coupled with a score of greater than or equal to 5 on a 7-point patient global impression of change scale.
Patient global impression of change (PGIC) score | 4 weeks
  1-7 scale evaluating, with higher scores indicating greater improvement.
Athens Insomnia Scale score | 4 weeks
  Scale measuring sleep dysfunction on an 8-question 0-24 scale, with higher numbers indicating greater dysfunction.
Hospital Anxiety and Depression Scale score | 4 weeks
  14-question scale measuring anxiety and depression, with each question scored as 0-3 (higher numbers represent greater anxiety or depression).
Pain pressure threshold | 4 weeks
  Pain pressure threshold, measured via algometry 3 times over the most tender area (mean of 3 measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - DC VA Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Blaustein Pain Treatment Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The protocol, and de-identified data may be shared with other researchers, pending approval (if relevant) from the Dept. of Defense (Walter Reed) and VA (DC VA Hospital)
Supporting Information: Study Protocol, Analytic Code
Time Frame: After publication, for at least 3 years
Access Criteria: Request, including objectives, to the Overall PI (SP Cohen)

REFERENCES:
- [Background] Predel HG, Giannetti B, Pabst H, Schaefer A, Hug AM, Burnett I. Efficacy and safety of diclofenac diethylamine 1.16% gel in acute neck pain: a randomized, double-blind, placebo-controlled study. BMC Musculoskelet Disord. 2013 Aug 21;14:250. doi: 10.1186/1471-2474-14-250. PMID 23964752
- [Result] Cohen SP, Hooten WM. Advances in the diagnosis and management of neck pain. BMJ. 2017 Aug 14;358:j3221. doi: 10.1136/bmj.j3221. PMID 28807894
- [Result] Hashmi JA, Baliki MN, Huang L, Parks EL, Chanda ML, Schnitzer T, Apkarian AV. Lidocaine patch (5%) is no more potent than placebo in treating chronic back pain when tested in a randomised double blind placebo controlled brain imaging study. Mol Pain. 2012 Apr 24;8:29. doi: 10.1186/1744-8069-8-29. PMID 22531485
- [Result] Lin YC, Kuan TS, Hsieh PC, Yen WJ, Chang WC, Chen SM. Therapeutic effects of lidocaine patch on myofascial pain syndrome of the upper trapezius: a randomized, double-blind, placebo-controlled study. Am J Phys Med Rehabil. 2012 Oct;91(10):871-82. doi: 10.1097/PHM.0b013e3182645d30. PMID 22854911
- [Result] Hsieh LF, Hong CZ, Chern SH, Chen CC. Efficacy and side effects of diclofenac patch in treatment of patients with myofascial pain syndrome of the upper trapezius. J Pain Symptom Manage. 2010 Jan;39(1):116-25. doi: 10.1016/j.jpainsymman.2009.05.016. Epub 2009 Oct 12. PMID 19822404